CLINICAL TRIAL: NCT05456568
Title: Investigating Value-Based Procurement and Patient Reported Outcomes From Adults With Lymphoedema Using a 12-week Home-based Programme of LymphAssistTM (Intermittent Pneumatic Compression)
Brief Title: LymphAssistTM at Home (LAAH)
Acronym: LAAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea Bay University Health Board (Other)
Collaborators: Lymphoedema Wales Clinical Network (Unknown); Swansea University (Other); Huntleigh Healthcare Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LymphAssist at home Protocol
Record Dates: First submitted 2022-06-21; First posted 2022-07-13 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Lymphedema Arm; Lymphedema of Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will use IPC daily at home for 12 weeks alongside usual and standard care
  Interventions: Device: LymphAssistTM Professional

INTERVENTIONS:
Device: LymphAssistTM Professional — An intermittent pneumatic compression (IPC) device that mimics manual lymphatic drainage. Participants use the device daily for 12 weeks alongside their usual and standard lymphoedema care
  Other Names: Hydroven 12

SUMMARY:
Lymphoedema is a life-long condition causing long-term swelling affecting people physically, mentally and socially. Daily self-management covers four main areas (skin care, activity / movement, compression and massage / light touch). Intensive clinic-based treatments are available alongside usual care, including intermittent pneumatic compression (IPC). Recent studies have explored the feasibility, acceptability and impact of home-based IPC. This study will further our understanding of home-based IPC in a Value-Based procurement study.

DETAILED DESCRIPTION:
Lymphoedema is a life-long condition causing long-term swelling. Lymphoedema mainly affects the extremities (arms / legs) and can occur at any age, affecting people physically, mentally and socially. Usual care focuses on life-long and daily self-management over four main areas (skin care, activity, compression and massage / light touch). Intensive clinic-based treatments are available alongside usual care. Intermittent pneumatic compression (IPC) helps move the lymph (fluid associated with the swelling) to offer comfort and reduce pain. Lymphoedema Services in Wales currently offer IPC in a clinic setting, despite reports suggesting that home use is helpful. To know more about this, this study will look to see if home use:

* Improves clinical and patient reported outcomes
* Is a good use of time and costs (efficient)
* Provides benefits that outweigh the cost of buying the IPC equipment

This study will recruit 40 patients with lymphoedema to use IPC daily at home for 12-weeks alongside their usual care. Information will be collected before and after the study including clinical measures (swelling, skin problems), patient reported outcomes (symptoms, quality of life) and experience. The study will compare the costs of procuring the IPC equipment with any benefits gained or costs avoided (less infections or hospital care). Participants will also be offered the chance to talk about their experiences of using IPC during an interview. Findings will be shared by publication and presentation. If the benefits are shown, lymphoedema services might be able to provide IPC for routine use at home through Value-Based procurement.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of lymphoedema (either primary or secondary) affecting lower or upper limbs
* Known to local lymphoedema services and receiving ongoing treatment for their lymphoedema
* Age 18 and over
* Able to given informed written consent
* Able to safely use the Pump, following written and / or verbal instruction in English or Welsh

Exclusion Criteria:

* Cognitive impairment / unable to safely use the Pump at home
* Truncal / root of extremity oedema
* Known or suspected deep vein thrombosis
* Known or suspected pulmonary embolism
* Thrombophlebitis
* Active or suspected cellulitis
* Severe peripheral neuropathy
* Uncontrolled or severe congestive heart failure
* Pulmonary oedema
* Ischaemic vascular disease
* Active cancer / metastases affecting the area of lymphoedema / undergoing cancer treatment
* Untreated ulcer / wounds
* Urinary of faecal incontinence (for patients with lower limb lymphoedema only)
* History of clostridium difficile
* Unable to communicate in English or Welsh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Changes in Lymphoedema-specific Patient Reported Outcome Measures using LYMPROM© | 0 days, 12 weeks
  The effect Intermittent Pneumatic Compression (IPC) has on Lymphoedema-specific Patient Reported Outcome Measure (LYMPROM©) scores. LYMPROM© is a lymphoedema specific PROM that captures 13 outcomes covering physical, social and emotional health domains. LYMPROM© version 1.2 (26/03/2021) uses a scale where patients can report each item using a 0-10 score, where zero represents no impact and 10 represents extreme impact. A higher score reflects a worse outcome. Four of the items also include a 'not applicable response' option. At the end of LYMPROM© there is a free text box for patients to report descriptively on any other impact.

SECONDARY OUTCOMES:
The feasibility of recruiting 40 participants over 18 months to a study using IPC at home using screening and recruitment logs | 0 days, 18 months
  Recruitment phases with no more than 15 participants recruited at a time will be reported, with a total of 40 participants recruited within the expected study time frame (18 months) as captured using the screening and recruitment logs.
The acceptability of using Intermittent Pneumatic Compression (IPC) at home for 12-weeks including self-reported use (frequency and dose) of IPC using participant completed diaries | 0 days, 12 weeks
  Participant compliance with daily use of IPC, as documented in the instruction manual, will be reviewed by self-report including the dose and frequency of IPC use as documented in the participant diary. Dose and frequency of use will be reported as percentages compared to protocol.
Changes in contacts with health and social care services before and after the study using the Use of health and social-service questionnaire Client Service Receipt Inventory (CSRI) | 0 days, 12 weeks
  Changes in access to health and social-service (primary and secondary care contacts frequency, mode of contact and health / social care professional seen) before and after the study.
Changes in recourse use within health and social care services before and after the study using the Use of health and social-service questionnaire Client Service Receipt Inventory (CSRI) | 0 days, 12 weeks
  Changes in use of prescribed treatment (prescribed medication, creams and dressings) before and after the study.
Changes in number of cellulitis episodes, hospital admissions (including length of stay), antibiotic use and number of days off work due to cellulitis as reported using the study case report form | 0 days, 12 weeks
  Number of cellulitis episodes before the study and cellulitis recurrence during the study, including hospital admissions and length of stay, antibiotic use and number of days off work due to cellulitis.
Changes in range of movement measures using the study case report form | 0 days, 12 weeks
  Range of movement will be assessed from 0 percent to 100 percent where a higher number indicates increased range of movement.
Changes in skin condition before and after the study including assessments of skin appearance (soft, fibrosis, discoloured) and the presence / absence of ulcers / wounds, Stemmer's signs and pitting oedema using the study case report form | 0 days, 12 weeks
  Skin appearance, texture and tests will be evaluated using standardised assessments as per the study case report form. All items are measured as the presence or absence of the condition with descriptors used to evaluate further.
Changes in excess limb volumes using LymcalcTM, which uses the cylindrical calculation for limb volume | 0 days, 12 weeks
  Limb volume is measured using standardised guidance within the study case report form (LymcalcTM which uses the cylindrical calculation). Using measurements taken at 4cm intervals for the affected and unaffected limb volumes are calculated and will be reported as changes from baseline to end of study (reported a mls and percent).
Changes in lymphoedema staging / severity using the International Society of Lymphology (ISL) Staging of Lymphoedema | 0 days, 12 weeks
  Lymphoedema staging / severity scales are not validated and none has achieved international agreement, therefore the ISL Staging of Lymphoedema will be reported alongside two other scales in use. The ISL has five stages; from 0 (a latent lymphoedema or sub-clinical phase where swelling is not yet evident) to stage III (where elephantiac changes are observed / marked skin changes). Stage 1 represents the accumulation of oedema / swelling and is reversible e.g. swelling will resolve upon elevation though there may be some pitting oedema. There are two stage II differentiated by the presence / absence of pitting oedema. Neither will resolve upon elevation and the absence of pitting marks an advanced / late stage of lymphoedema with excess subcutaneous fat / fibrosis developing.
Changes in lymphoedema staging / severity using the British Lymphology Society (BLS) Grouping of Lymphoedema | 0 days, 12 weeks
  Lymphoedema staging / severity scales are not validated and none has achieved international agreement, therefore the BLS Group of Lymphoedema will be reported alongside two other scales in use. The BLS Groups begin with zero (a latent but high risk of lymphoedema phase) to stage four (palliative / end of life). Group one represents early lymphoedema (present for less than three months) where the swelling may resolve upon elevation for example. Group two represents established uncomplicated lymphoedema which no longer resolves upon elevation. Group three reflects complex lymphoedema with skin changes. There are three further sub categories within group three differentiated by the number of limbs affected or the presence of midline lymphoedema.
Changes in lymphoedema staging / severity using the Lymphoedema Wales Clinical Network (LWCN) Lymphoedema Severity Outcomes of Lymphoedema | 0 days, 12 weeks
  Lymphoedema staging / severity scales are not validated and none has achieved international agreement, therefore the LWCN Lymphoedema Severity Outcomes are reported alongside two other scales in use. This scale starts at one (at risk of lymphoedema but with no swelling at present). Outcome two represents mild lymphoedema with 5-10% difference in volumes (between affected and unaffected limbs). Outcome three represents moderate lymphoedema with 10-20% volume difference and four represents severe lymphoedema (21-49% volume difference). The final outcome is group five which has a further sub category to indicate the presence of a wound. Outcome five represents complex lymphoedema (more than or equal to 50% volume difference). This is the only scale to report separately on the presence of wounds.
Changes in health-related quality of life using the EQ-5D-5L | 0 days, 12 weeks
  Changes in quality of life scores and quality adjusted life years Health-related quality of life will be measured using the five-level EuroQol Five Dimensions (EQ-5D-5L). It is a non-disease specific tool to report health-related quality of life. The EQ-5D-5L includes five dimensions and a visual analogue scale (EQ-VAS). Each of the five dimensions are each reported with five responses (from no problems, slight problems, moderate problems, severe problems, and extreme problems). The five dimensions are mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. For each of the five dimensions a 5-digit health state profile can be produced. The VAS records self-perceived health on the present day using a vertical thermometer from 0 (worst imaginable health) to 100 (best imaginable health).
Changes in work and activity as reported using the Work Productivity and Activity Impairment Questionnaire: Lymphoedema (WPAI-Lymphoedema) | 0 days, 12 weeks
  WPAI has six items, the first is a dichotomous item to denote if the individual is in paid employment. The remainder of items are used to report presenteeism / absenteeism, productive loss and activity impairment. WPAI: Lymphoedema scores are presented as percentages where higher numbers indicate greater impairment and less productivity.
Procurement and life-time costs of home use compared with clinic based treatment | 0 days, 12 weeks
  The purchase (procurement) costs will be reported and evaluated alongside direct and indirect healthcare costs using the Client Service Receipt Inventory (CSRI) - outcome three. Ongoing costs (clinician time) for home versus clinic-based IPC use will be reported in pound sterling (GBP).
Number of participants with treatment-related adverse events and their severity and relationship to the study as assessed by Participant Adverse Event Log | 0 days, 12 weeks
  Number and nature of problems found when using IPC for 12-weeks at home will be reported using the Participant Adverse Event Log. This will include reporting on the severity, likelihood and relationship to study treatment.
Attrition will be reported in terms of number of participants recorded as loss to follow up as captured in the case report forms and study flow diagram. | 0 days, 18 months
  Loss to follow-up of participants will be enumerated and described where reasons are provided as captured in the case report forms and reported in the study flow diagram.

OTHER OUTCOMES:
Patient experience | 12 weeks
  An interview guide has been developed for the semi-structure interviews covering: living with lymphoedema; experiences of lymphoedema management and Intermittent Pneumatic Compress (IPC) at home.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Gabe-Walters, PhD, Principal Investigator — Lymphoedema Wales
Locations (1):
- Swansea Bay University Health Board, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No